CLINICAL TRIAL: NCT05761717
Title: Clinical Study of mRNA Personalized Tumor Vaccine Encoding Neonatal Antigen Combined With Sintilimab Injection Liver Cancer
Brief Title: Clinical Study of mRNA Vaccine in Patients With Liver Cancer After Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-10-mRNA-COM
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Posto Perative Hepatocellular Carcinoma

STUDY DESIGN:
Intervention Model Description: 12~18 participants in Cohort . C1:50 ug of PCV; C2: 100 ug of PCV ; C3: 150 ug of PCV.Extended research phase:49 participants in Cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3+3 (Experimental): Neoantigen mRNA Personalised Cancer in combination with Stintilimab Injection. This study is a 3+3 dose escalation design.Participants will receive a total of 6 cycles of PCV every 21 days
  Interventions: Drug: Neoantigen mRNA Personalised Cancer vaccine in combination with Stintilimab I njection

INTERVENTIONS:
Drug: Neoantigen mRNA Personalised Cancer vaccine in combination with Stintilimab I njection — Subcutaneous Injection

SUMMARY:
This is an open, one-arm study to evaluate the safety and efficacy of mRNA personalized tumor vaccine (tumor vaccine) encoding neonatal antigen in combination with Sintilimab injection for adjuvant prevention of postoperative recurrence of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥18 years old (including boundary values), without limitation of sex at time of consent.
* The patient was confirmed as hepatocellular carcinoma by histopathology or cytology after surgery, and the lesion was completely resected by surgery R0 (no residual tumor under postoperative microscope and naked eye), and no residual lesion or extrahepatic metastasis was confirmed by postoperative imaging (CT/MRI).
* The patient is at high risk of postoperative recurrence, and the tumor must meet the following characteristics: Patients with hepatocellular carcinoma IIb/IIIa as defined by the 2019 Chinese Staging System.
* The Eastern Oncology Consortium Physical State Score (ECOG PS) is 0 or 1, and the Child-Pugh rating is A

Exclusion Criteria:

* Known allergy to any tumor vaccine, adjuvant, Stintilimab Injection formulation, fluorouracil inj, oxaliplatin injcalcies;
* Tumor mutation load (TMB) was less than 2.0/Mb or neonatal antigen load (TNB) was less than 0.5/Mb or the predicted number of neonatal antigens was less than 15;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2025-03-12 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
One-year recurrence-free survival rate (RFS); | 1 year
Overall survival (OS) after initial administration. | 1 year